CLINICAL TRIAL: NCT04752917
Title: Do Noise Cancelling Headphones Reduce Patient Controlled Midazolam Requirements in Primary Knee Arthroplasty Patients Under Spinal Anaesthesia
Brief Title: Do Noise Cancelling Headphones Reduce Sedation Requirements in Primary Knee Arthoplasty
Acronym: NOISE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Chief Investigator retirement
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STH20161
Record Dates: First submitted 2019-08-29; First posted 2021-02-12 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Anaesthesia; Knee Surgery

STUDY DESIGN:
Intervention Model Description: Randomised trial of control and intervention groups
Who Masked: Participant
Masking Description: Unblinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Headphones
  Interventions: Device: Noise Cancelling headphones
- Control (No Intervention): Standard of care

INTERVENTIONS:
Device: Noise Cancelling headphones — Use of headphones playing patients choice of music
  Arms: Intervention

SUMMARY:
The study is a randomised trial of headphones with midazolam patient controlled sedation (intervention group) vs control group with no heaphones to compare sedation usage during knee replacement surgery under spinal.

The trial is a pilot study of 20 cases

DETAILED DESCRIPTION:
The study is for patients undergoing elective primary knee replacement surgery under spinal anaesthesia. It is proposed that using music played on noise cancelling headphones will reduce the requirements for intravenous sedation in a randomised controlled trial of twenty patients. Spinal anaesthesia is commonly used for knee replacement. It provides loss of feeling from the operated limb but the patient remains awake. Orthopaedic surgery is very noisy. It is usual for patients to receive intravenous sedation with midazolam to reduce their awareness of surgery. Intravenous midazolam is effective but it depresses both the breathing and the circulation and may cause low blood pressure and reduced oxygenation. It is expected that by using noise cancelling headphones to reduce the awareness of noise during surgery, there will be a reduced requirement for intravenous midazolam. The study will measure the dose of midazolam required by patients randomised to receive either noise cancelling headphones playing music (intervention) or no headphones (control group). Patients will be followed up prior to hospital discharge to assess their awareness and recall of intra operative events and their satisfaction with intravenous sedation. This is a novel application of sound reducing technology capable of improving the patient experience during surgery whilst potentially reducing complications of intravenous midazolam sedation. Noise cancelling technology is readily available in commercially available headphones and it has the potential to eliminate background noise of surgical procedures. This study findings will be of interest for health professionals and patients involved in surgery or investigative procedures normally carried out with intravenous sedation.

ELIGIBILITY:
Inclusion Criteria:

* Elective primary knee surgery under spinal anaesthesia
* Willing to receive patient controlled midazolam sedation

Exclusion Criteria:

* Deafness
* Unwilling to use headphones
* Unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2021-08-24 (Actual)

PRIMARY OUTCOMES:
Change of sedation requirements during elective orthopaedic surgery. | 3 hours
  Measuring the difference in intravenous sedation requirements for patient controlled midazolam during elective primary knee joint replacement surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Marks, Dr, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
This is pilot data and will hopefully lead to an application for a larger definitive study